CLINICAL TRIAL: NCT02185287
Title: "The Urological Dysfunctions in Young Women: Inheritance of Childhood?"
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Collaborators: University Of Perugia (Other)
Responsible Party: Principal Investigator, Antonio Luigi Pastore, Assistant Professor, MD, PhD, University of Roma La Sapienza
Other Study IDs: 2199/13 Prot.N.1625/13/ON
Record Dates: First submitted 2014-07-01; First posted 2014-07-09 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Lower Urinary Tract Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lower urinary tract dysfunction, female, age: 18-40 years
- Healthy female subjects, age: 18-40 years

SUMMARY:
Aim of the study protocol is to evaluate in a prospective investigation of health statistics if the dysfunctions of the lower urinary tract in women aged between 18 and 40 years may be the result of past urinary pediatric dysfunction. The aim is to be able to identify the "risk conditions" which, if treated properly in early childhood, to help avoid debilitating problems that manifest themselves as adults and possibly to implement a strategy of prevention.

The choice of this age group is due to the fact that it allows for easier retrieval of data, as it is presumed that the concerned can more easily remember their history of pediatric and / or have parents still young enough to ask for such information. The problems of urinary disorders in childhood era have been the subject of increased attention by pediatricians from the end of the 70s, therefore, history taking may be more complete.

A study by Fitzgerald evaluated female subjects with mean age of 56 ± 9 years, and therefore our study aim is to investigate an age group that does not appear in the literature to supplement these findings, already reported.

Ultimate goal is the need to raise awareness of Pediatric Urologists to interact with adult Urologists in order to implement a shared strategy for the management of patients with problems of impaired bladder function in order to improve the future lower urinary tract function.

Materials and Methods: A self administered questionnaire will be used in accordance with the guidelines of the International Children's Continence Society. The questionnaire consists of two parts: the first explores the history of urological clinic patient until the age of 14,in order to evaluate any symptoms reported in a specific category of typical dysfunction of childhood; the second part refers to the present together with urological disorders of sexual function which, as emerges from the data of the literature may be of relevance urological diseases detectors. The data obtained will then be subjected to statistical calculations by which will evaluate the significance of the symptoms present in childhood in relation to their penetrance in various forms of adult diseases dysfunctional bladder and / or sexual abuse, with the prediction of the evolution of the same.

The questionnaire is anonymous in order to protect privacy. The questions that comprise it have been partly extracted from the questionnaire validated by the International Children's Society Continent and partly made by the authors of this study on the basis of the scientific evidence.

Patients will be recruited from the outpatient clinic of the Urogynecology Urology Clinic, University of Perugia, while the healthy controls will be recruited by submitting a questionnaire to the women chosen to sample a healthy population of Graduate Schools found in the framework of Urology, Pediatrics and Pediatric Surgery, University of Perugia.

The Investigators defined that the statistically significant number of healthy and pathological subjects can not be less than 200 units per reference category.

The time duration of the collection of anamnestic data depend on the ability of the authors of this research in finding the subjects to be analyzed.

There are no conflicts of interest to declare, no drugs or medical equipment will be tested .

ELIGIBILITY:
Inclusion Criteria:

* Any lower urinary tract symptoms
* Female aged between 18 and 40 years

Exclusion Criteria:

* Age limit
* Lower urinary tract infection

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients will be recruited from the outpatient clinic of the Urogynecology Urology Clinic, University of Perugia, while the healthy controls will be recruited by submitting a questionnaire to the women chosen to sample a healthy population of Graduate Schools found in the framework of Urology, Pediatrics and Pediatric Surgery, University of Perugia.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
International Children Continence Society Questionnaire | Questionnaires scores at time 0 (screening time)

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Urology Unit, Sapienza University of Rome, Latina
  - Pediatric Surgery, University of Perugia, Perugia
  - Urogynecology Unit, Urology Clinic, University of Perugia, Perugia

REFERENCES:
- [Background] Kuh D, Cardozo L, Hardy R. Urinary incontinence in middle aged women: childhood enuresis and other lifetime risk factors in a British prospective cohort. J Epidemiol Community Health. 1999 Aug;53(8):453-8. doi: 10.1136/jech.53.8.453. PMID 10562862
- [Background] Fitzgerald MP, Thom DH, Wassel-Fyr C, Subak L, Brubaker L, Van Den Eeden SK, Brown JS; Reproductive Risks for Incontinence Study at Kaiser Research Group. Childhood urinary symptoms predict adult overactive bladder symptoms. J Urol. 2006 Mar;175(3 Pt 1):989-93. doi: 10.1016/S0022-5347(05)00416-7. PMID 16469599
- [Background] Falconer C, Ekman-Ordeberg G, Hilliges M, Johansson O. Decreased innervation of the paraurethral epithelium in stress urinary incontinent women. Eur J Obstet Gynecol Reprod Biol. 1997 Apr;72(2):195-8. doi: 10.1016/s0301-2115(96)02685-1. PMID 9134401